CLINICAL TRIAL: NCT04323215
Title: One Year Evaluation of a Web-based System for Optimization of Behavioural Childhood Obesity Treatment
Brief Title: Evaluation of a Digital Childhood Obesity Treatment
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal Investigator, Karolinska Institutet
Other Study IDs: Provement100
Record Dates: First submitted 2020-03-17; First posted 2020-03-26 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity; Treatment Adherence
Keywords: Mobile Health; Support System; Behavioral treatment; Self-Monitoring
MeSH Terms: conditions — Pediatric Obesity; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Support system users: Usual care (behavioral treatment) plus the support system for self-monitoring of weight and communication with the clinic during one year of treatment.
  Interventions: Device: Support system
- Control group: Children treated with usual care according to regular treatment routines registred in BORIS the Swedish childhood obesity treatment register

INTERVENTIONS:
Device: Support system — A support system named Provement will be used to provide behavioral treatment.
  Groups: Support system users

SUMMARY:
This study aims to evaluate if a web-based digital support system aiming to replacing or complement standardized pediatric behavioural obesity treatment. The hypothesis is that a digital system of communication between the family and the clinic can generate improved treatment results (change in BMI SDS) and reduce the number of missed visits.

DETAILED DESCRIPTION:
Childhood obesity treatment is time consuming for both the health care system, and for the involved families. There is an association between the intensity and the outcome of treatment.

In this study all children who start treatment for childhood obesity will use a digital support system as a complement to behavioral treatment. The digital support system includes daily weighing on scales that do not show any digits, linked to a mobile app where weight development is shown as a moving average in the form of BMI standard deviation score (SDS). The app also provides an individual target curve visualizing the expected weight journey. Weight in growing children is complex to interpret why BMI SDS is used. Objective data from scale are automatically transferred to the database and the clinic and the family have direct contact with the clinic via the app.

The evaluation will be carried out when approximately 120 children have had the opportunity to be treated with the support system for one year. The results will be compared with a matched control group from the BORIS childhood obesity treatment register.

ELIGIBILITY:
Inclusion Criteria:

* Obesity according to International Obesity Task Force (IOTF)

Exclusion Criteria:

* No

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children who start treatment for childhood obesity at Martina children Hospital will use a digital support system as a complement to behavioral treatment. Approximately 120 children 3-18 years will be included in this first evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in degree of obesity | From start of treatment to one year follow-up
  Measured by BMI standard deviation score. Support system users vs control

SECONDARY OUTCOMES:
The use of the support system - weighings | From start of treatment to one year follow-up
  Number of weighings/week
The use of the support system - text messages | From start of treatment to one year follow-up
  Number text messages/week
Number of physical visits | From start of treatment to one year follow-up
  Visits to the clinic. Support system users vs control
Number of cancelation of physical visits | From start of treatment to one year follow-up
  Visits to the clinic. Support system users vs control
Number of patients not showing up to physical visit | From start of treatment to one year follow-up
  Visits to the clinic. Support system users vs control

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet, CLINTEC, Division of pediatrics
Locations (1):
- Childrens hospital Martina, Stockholm, Sweden

REFERENCES:
- [Derived] Hagman E, Johansson L, Kollin C, Marcus E, Drangel A, Marcus L, Marcus C, Danielsson P. Effect of an interactive mobile health support system and daily weight measurements for pediatric obesity treatment, a 1-year pragmatical clinical trial. Int J Obes (Lond). 2022 Aug;46(8):1527-1533. doi: 10.1038/s41366-022-01146-8. Epub 2022 May 31. PMID 35641569